CLINICAL TRIAL: NCT03981458
Title: Hyaluronate for the Treatment and Prevention of Recurrent Urinary Tract Infection in Women Suffering Atrophic Vaginitis
Acronym: HATPIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: The Urology Foundation, UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HATPIN; 8904 (Other: R&D Number Newcastle Hospitals)
Record Dates: First submitted 2019-01-29; First posted 2019-06-10 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Atrophic Vaginitis; Urinary Tract Infections
MeSH Terms: conditions — Atrophic Vaginitis; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Atrophic vaginitis and recurrent urinary tract infection are often found concurrently in post-menopausal women. The argument over which condition appeared first, or if one is caused by the other, is prevalent in clinical settings and there is no official guidance as to which should be treated first. We propose two arms to this study - one treating the atrophic vaginitis via use of Hyalofemme cream (hyaluronate cream), and the other treating recurrent UTI by use of Ialuril (hyaluronate bladder instillation). We intend to investigate the effect on the incidence of UTI in the patients with both treatments, as well as focusing on some markers of the immune response in the urine and vaginal douche samples from these participants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyalofemme (Active Comparator): Hyalofemme is a cream/gel containing hyaluronic acid, designed to be applied vaginally. This is primarily used in treatment of atrophic vaginitis and is applied by the patient once every three days. We intend treatment to continue for 6 months.
  Interventions: Device: Hyalofemme
- Ialuril (Active Comparator): Ialuril is a bladder instillation designed to be delivered to the bladder via catheter. This is primarily used in patients suffering from recurrent UTI and acts to help rebuild the lining of the bladder, reducing irritation. Ialuril is applied weekly for 6 weeks, followed by every 2 weeks for 6 weeks, then once monthly for maintenance. Treatment will be continued for 6 months.
  Interventions: Device: Ialuril

INTERVENTIONS:
Device: Hyalofemme — Gel made with hyaluronic acid to be applied vaginally to treat atrophic vaginitis.
  Other Names: Hyaluronic acid gel; Hyaluronate gel
  Arms: Hyalofemme
Device: Ialuril — Bladder instillation of hyaluronic acid to treat recurrent UTI.
  Other Names: Hyaluronic acid instillation; Hyaluronate instillation
  Arms: Ialuril

SUMMARY:
In post-menopausal women, the condition atrophic vaginitis results from the loss of oestrogen and is characterised by dyspareunia (pain during intercourse), vaginal dryness, and vaginal irritation. It is often diagnosed alongside recurrent urinary tract infections (rUTIs) and may increase susceptibility to rUTI. Topical vaginal oestrogen can be used to re-condition the vaginal epithelium and also reduces the incidence of rUTIs. However, patients often express concerns about using oestrogen, a hormonal treatment. Studies also report side-effects including vaginal bleeding, discharge, burning and itching that underpin significant (28%) drop-out rates. Hence, alternative non-hormonal, non-antibiotic based therapies that treat the vaginal atrophy, but also reduce the incidence of rUTI are needed.

Recurrent UTI in adult women is common. Bacteria from the gut can colonise the vulvar epithelia and then the bladder, causing uncomfortable urinary symptoms (cystitis). The lifetime risk of a UTI is around 40% in adult women which increases in post-menopausal women. Annually, UTI incidence is 3%. Of those affected, 5% will suffer rUTI, rising to 13% in the over 60 population. This equates to over 300,000 of the adult female UK population annually affected by rUTI. The most frequent treatment for rUTIs is low dose antibiotics, but this treatment causes the bacteria carried by such women to become antibiotic resistant, which exacerbates the clinical problem. The prevalence of antimicrobial multi-resistance within post-menopausal women suffering from rUTI is around 25% and was shown to rise to more than 80% following prolonged antibiotics. These data support the use of non-antibiotic treatment strategies that prevent rUTI and the emergence of drug resistant micro-organisms.

This study will compare two groups with differing treatment strategies. One group will be primarily treated for atrophic vaginitis with topical vaginal hyaluronate and the other will be primarily treated for their recurrent UTI with intravesical hyaluronate.

DETAILED DESCRIPTION:
Study purpose A potential alternative to prophylactic antibiotic treatment and topical vaginal estrogen treatments is the compound hyaluronate (HA). HA is already utilised in the UK to treat rUTIs, but is delivered as a bladder instillation (Ialuril®). A small meta-analysis of intravesical hyaluronate therapy incorporating four studies (two randomised, two non-randomised, 143 patients) investigating the use of this treatment in recurrent UTI, reported a statistically significant improvement in the rates of recurrent UTI (mean difference -3.4 episodes per patient year, 95% confidence interval -4.3 to -2.5). HA is also available as a vaginal cream, Hyalofemme®, which is used clinically to treat atrophic vaginitis. The evidence suggests that many women suffering vaginal atrophy also experience recurrent UTIs. However, the effect of HA treatment in reducing concomitant rUTIs in such patients has not been reported.

The need for this study is also supported by current guidance documents. The 2012 Scottish Intercollegiate Guideline Network (SIGN) guideline emphasises the need to avoid "unnecessary antibiotic prescribing," specifically highlighting the issue of antibiotic-resistant [E. coli] UTI. Additionally, the UK antimicrobial resistance strategy documents antibiotic resistance as a key concern and as such, lends support to the investigation, and use of alternative antimicrobial therapies. The use of non-antibiotic preventative treatments for rUTI has also been accentuated by current UK, European and USA guidelines to minimise antibiotic resistance. Therefore, this pilot study investigating the efficacy of a treatment already prescribed for vaginal atrophy in reducing concomitant rUTI is not only addressing current directives, but will help inform whether topical HA therapy can be extended to all rUTI sufferers, thus helping to reduce global antibiotic use.

Evidence supporting the effectiveness of hyaluronate (HA) in treating rUTI is available, but at present the therapy is administered directly to the bladder, which involves catheterisation, managed through hospital visits. In contrast a HA topical treatment can be patient managed at home. If from the data collated the topical HA therapy shows a comparable efficacy in reducing rUTI, then these data will underpin a large-scale clinical trial examining the use of this non-hormonal, non-antibiotic based agent for the treatment and prevention of rUTI in patients.

While the focus of this initial study is on post-menopausal women suffering vaginal atrophy and rUTI, it is also anticipated that this treatment could be broadened to all women suffering rUTIs. One particular target group are females carrying the TLR5392Stop polymorphism who are at increased risk of rUTI, thus signalling an era of personalised medicine for an infection related disease. It is also envisaged that topical HA therapy could be prescribed as a urethral barrier cream for men suffering uncomplicated rUTI.

Study design This study was designed through a collaboration of clinical urologists and basic scientists with an interest in the concomitance of atrophic vaginitis and recurrent UTI. The proposal was peer-reviewed before funding was granted by The Urology Foundation. This single-centre study is located at the Urology Department, Freeman Hospital, Newcastle upon Tyne Hospitals NHS Foundation Trust, NE7 7DN. Participants recruited will be post-menopausal women identified as either having gone through the menopause naturally or having had an oophorectomy, and not on hormone replacement therapy (HRT) in the last two years, and who suffer from vaginal atrophy and rUTI. Patients will have either 3 confirmed episodes of UTI in the preceding year or 2 episodes in the last 6 months. Patients will exhibit the symptoms and signs of atrophic vaginitis, which will be diagnosed by their responsible clinician. The study duration is 24 months, with a patient recruitment period of 12 months. Patient follow up and laboratory work will proceed until the end of month 23, with data analyses and final report preparation in the final month.

The design incorporates a patient-randomised study that directly compares two treatments for women with atrophic vaginitis and rUTI during a 9-month period. One treatment is an intravesical instillation of hyaluronate into the bladder (Ialuril) delivered via catheter focussed primarily on treating rUTI. This is once weekly for 6 weeks, followed by once every two weeks for 6 weeks, then once per month (maintenance) for the remaining study period. The alternative treatment is focussed on primarily treating atrophic vaginitis using a licensed vaginal hyaluronate product (Hyalofemme) used topically once every 3 days, continually for the 9 month study period.

Participants in both study arms would continue to receive antibiotic treatment for breakthrough UTI as needed. Recruitment is planned at 3-4 patients per month, allowing us to meet a target of 40 participants over the recruitment period, which allows for a 25% attrition rate. Using data from Damiano et al, two groups of 16 patients are required to achieve 80% power at the 5% significance level for detecting a clinically significant reduction of one less UTI during the 9-month treatment and monitoring period.

Recruitment

1. Patient Identification All adult women with atrophic vaginitis and rUTI will be made aware of the study during their clinic appointment and those eligible can consider whether they wish to participate prior to assessment. The study will also be publicised so that colleagues in allied specialities such as urogynaecology and nephrology, who may receive referrals of women with atrophic vaginitis and rUTI, are aware of the study and can identify potential participants.

   For the study, post-menopausal women with symptoms or signs of atrophic vaginitis referred to a hospital urology clinic with associated rUTI will be asked if they would like to participate. In the study, atrophic vaginitis will be diagnosed on clinical grounds and rUTI will be defined as at least 3 episodes in the past year (or 2 episodes in the last 6 months). Patients will undergo routine tests to rule out any structural or functional abnormality of their urinary system. The treatment given to each participant will be decided randomly.

   Patients with underlying structural or functional abnormalities of the urinary tract following diagnosis by renal tract ultrasound scan (USS) and an endoscopic examination of the bladder under local anaesthesia (flexible cystoscopy) will be excluded from the study. A recent local audit in Newcastle (unpublished data, n=200) has revealed that contributory structural or functional abnormalities are detected in less than 10% of patients. Therefore, it is estimated that approximately 90% of patients matching our criteria and referred with atrophic vaginitis and rUTI will be eligible to be approached for inclusion to the study.

   Recruitment will involve a clear explanation of the trial including the background, study protocol and aims.
2. Screening Clinical staff at each site will identify eligible participants through direct contact or by searches of electronic records held in each Trust. They will then give or send potentially eligible patients brief study information. If interested potential participants can then agree to be approached by research staff and be provided with further study information. Invitation material will include brief details of the need and purpose of the study and eligibility criteria. It will emphasise the pragmatic nature of the study and give a realistic indication of the burden to participants. All patients given study information will be recorded in the screening log. All subjects who agree to consider participation will be seen by local research staff or the study coordinator to go through the consent and randomisation procedure. A case report form will be initiated and baseline data collected.

   A screening log will be kept by local site research staff to document details of subjects invited to participate in the study and reasons for non-participation. The log will also ensure potential participants who are ineligible or decline participation are approached only once.
3. Consent All participants will undergo a process of informed consent. Participants will be free to withdraw their consent at any time.

The informed consent discussion will be undertaken by appropriately trained staff. This will include medical staff and research nurses/study coordinators involved in the study who will give time for participants to ask any questions they may have following review of the study information pack. The consent process will include written information concerning the need and overall benefit of the study as well as verbal discussions. The latter will include a check of understanding concerning benefits and risks, and ensuring that participants accept that the treatment will be allocated at random regardless of any personal preference they may have.

Following delivery of the study information, participants will be given at least 24 hours and as much time as they need to decide whether they would like to participate. Those wishing to take part will provide written informed consent by signing and dating the study consent form, which will be witnessed and dated by a member of the research team with documented, delegated responsibility to do so. Written informed consent will always be obtained prior to randomisation. The original signed consent form will be retained in the Investigator Site File, with a copy filed in the clinical notes, a copy given to the participant. The participant will specifically consent to their General Practitioner (GP) being informed of their participation in the study. The right to refuse to participate without giving reasons will be respected.

Participants will be given the option of consenting to storage of blood, urine and vaginal douche samples for future research. They will also be asked if they would be willing for the inclusion of data collected for this study in future research. Any further research would be subject to separate review by an ethics committee.

Inclusion/exclusion and risk Selection bias will be minimised by including all post-menopausal female patients with atrophic vaginitis and recurrent uncomplicated UTI, and not receiving hormonal supplements or hyaluronate as eligible participants. There are deliberately few exclusion criteria set to enable the findings of this study to be generalised. Both treatments are licensed, exhibit a low side-effect profile and have little interaction with other common medications, which limits absolute contra-indications to either therapy. Eligible patients and their responsible clinician will need to be sufficiently uncertain of the optimum treatment for vaginal atrophy and rUTI to allow randomisation and prevent selection bias.

Confidentiality Initial screening of patients will be carried out by trained clinical staff associated with either the urology clinic at Freeman Hospital or the network of Research Nurses. Following this, informed consent will be taken by appropriately trained staff and the patients randomised into the trial. Case Report Forms to collect the information required by researchers will contain the minimum required patient-identifiers. All staff have completed GDPR training.

Conflict of interest This study is pragmatic in design and, apart from random allocation of treatment option and participant completion of diaries and questionnaires, participant care will follow standard pathways in participating secondary care NHS sites. Both Ialuril and Hyalofemme are licensed and approved for routine NHS use. It will be ensured that all participants have access as desired to the use of other measures to reduce the risk of UTI such as adequate fluid intake, avoidance of constipation and cranberry extract. However, patients receiving hormonal supplementation are not appropriate for this study. Participants in both study groups will receive on demand discrete courses of antibiotics as decided by the responsible clinician for symptomatic UTI. Use of all these adjunctive treatments will be recorded on case report forms.

Participants will be given the option of consenting to storage of blood, urine and vaginal douche samples for future research. Participants will also be asked if they would be willing for the inclusion of data collected for this study in future research. Any further research would be subject to separate review by an ethics committee. Upon completion a short, clearly written summary of the research findings will be supplied to all participants. Any findings resulting from the research will be published in scientific or medical journals.

ELIGIBILITY:
Inclusion Criteria:

* • Postmenopausal women not receiving hormonal supplementation.

  * Women with atrophic vaginitis and rUTI who, in consultation with a clinician, have decided that either hyaluronate treatment (intravesical or vaginal) is an appropriate option.
  * Women who have suffered at least three episodes of symptomatic UTI within the preceding 12 months or two episodes in the last 6 months.
  * Able to attend a urology clinic for catheterisation on a regular basis (initially weekly) to initiate intravesical bladder instillation treatment.
  * Able to apply vaginal hyaluronate gel at home every 3 days.
  * Able to give informed consent for participation in study.
  * Able and willing to adhere to a 9-month study period.

Exclusion Criteria:

* • Postmenopausal women receiving hormonal supplementation (e.g. HRT or oestrogen creams).

  * Women unable to use hyaluronate e.g. due to previous sensitivity issues.
  * Women with urinary tract abnormalities that are considered to be contributory to the occurrence of rUTI.
  * Presence of symptomatic UTI - this will be treated and symptoms resolved prior to randomisation.
  * Women currently using hyaluronate for either treatment of atrophic vaginitis or prevention of recurrent UTI or women who have used either study treatment in the preceding 12 months.
  * Women receiving prophylactic antibiotics.
  * Catheter usage.

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Reduced incidence of medically confirmed urinary tract infection | Number of UTIs will be assessed at both 6 months (end of treatment) and 9 months (end of follow-up period)
  Occurrence of symptomatic UTI with prescription and taking of a treatment course of antibiotics for UTI. Applicable for both treatment arms in comparison to baseline established in the previous 12 months.

SECONDARY OUTCOMES:
Number of microbiologically-proven UTIs | 6 and 9 months
  Occurrence of symptomatic UTI and the demonstration of a positive urine culture, rather than UTI symptoms potentially caused by interstitial cystitis without bacterial infection.
Effect on vaginal atrophy | 3, 6 and 9 months
  The two treatment arms will be compared to baseline to discover whether any improvement in vaginal atrophy symptoms are seen with either treatment. This will be assessed via questionnaires to determine symptoms experienced and their severity at 0 (baseline), 3, 6 and 9 months. Symptoms that participants will be asked to assess are as follows:
  * Frequency of urination
  * Urgency of urination
  * Pain or burning during urination
  * Partial bladder emptying
  * Fever or shivers
  * Pain in the lower abdomen or pelvis
  * Lower back pain
  * Blood in the urine Participants will rank the severity of these symptoms from "Did not have" to "Severe", and how troublesome they were from "Not at all" to "A lot" by marking a line to indicate where the participant feels their symptoms lie. Upon analysis of the questionnaires, placement of this mark will be measured and used to determine differences in symptoms from baseline throughout the study.
Uropathogen identification | 9 months
  Urine samples will be analysed for the presence of bacteria. If any are found they will be cultured, identified and potentially undergo molecular typing to discover whether particular strains are more prevalent in patients suffering from concurrent rUTI and atrophic vaginitis.
Innate immune response in urine and vaginal douche samples measured by ELISA for cytokines and antimicrobial peptides (e.g. interleukin-8, beta-defensin 2). | 9 months
  Urine and vaginal douche samples will be collected at baseline and at 3-monthly intervals. These will be analysed by ELISA for the presence of innate immune markers and cytokines, such as defensins, interleukin-8 and lipocalin. A potential change in expression may indicate that this is partly how the treatments help to prevent against UTI.
Analysis of polymorphisms in receptor proteins known to be involved in UTI | 9 months
  Patient blood samples will be collected at baseline and DNA extracted. These will be examined for SNPs in genes such as TLR5, which encodes a receptor protein known to affect patient response to bacteria in cases of UTI.
Participant quality of life - does either treatment increase overall quality of life by decreasing symptoms from UTI and/or atrophy? | 3, 6 and 9 months
  Participants will be asked to complete questionnaires (EQ-5D) pertaining to their overall health and quality of life at baseline and at 3-monthly intervals to determine whether treatments are improving their overall health and general wellbeing at 0, 3, 6 and 9 months. This is a validated questionnaire commonly used in healthcare to determine general health and includes assessments of mobility, self-care, ability to carry out normal activity, pain/discomfort levels and anxiety/depression. This also asks participants to assess their overall health state by marking on a scale from 0-100, with higher numbers representing the best imaginable state of health.
Reduction in antibiotic use for UTI as a result of hyaluronate treatment by either route of administration | Results will be analysed at both end of treatment (6 months) and end of follow-up (9 months)
  Incidences of antibiotic use, in general and specifically for UTI, will be recorded to observe whether the treatments result in fewer courses of antibiotics being prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Harding, MD, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No